CLINICAL TRIAL: NCT02483325
Title: Phase II Study Evaluating the Efficacy of Allogeneic Transplant Conditioning With Adaptive Dose Busulfan Intravenous (Busilvex®) in Patients at High Risk of Carrying Blood Diseases
Brief Title: Study Evaluating the Efficacy of Allogeneic Transplant Conditioning With Adaptive Dose Busulfan Intravenous (Busilvex®) in Patients at High Risk of Carrying Blood Diseases
Acronym: BX-PK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BX-PK-IPC 2013-016
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Hematological Diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Busulfan; Antilymphocyte Serum; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Busulfan with adapted doses (Other): Conditioning regimen for allogeneic transplant (Busulfan, Thymoglobuline and Fludarabine)
  Interventions: Drug: Allogeneic transplant conditioning

INTERVENTIONS:
Drug: Allogeneic transplant conditioning — Allogeneic transplant
  Other Names: Busulfan, thymoglobuline, fludarabine

SUMMARY:
Determine the efficiency of a myéloablative conditioning associating Fludarabine, Thymoglobuline, and intravenous Busulfan with adapted dose, according to a pharmacokinetics realized in the first day of administration (or J-6 of the conditioning) of the busulfan, in preparation for a allogenic transplant family or not family compatible HLA.

ELIGIBILITY:
Inclusion Criteria :

* Informed consent signed,
* Patient affiliated to a social security system or benefiting from such a system,
* Related HLA identical donor or unrelated HLA identical donor :

all patients aged > 55 years with hematological malignancy and deemed eligible for an allogeneic transplant from a geno-identical donor and pheno-identical 10/10

- the basic pathology should be considered "chemo-sensitive" complete or partial remission (CR, PR) or stable disease

Exclusion Criteria :

* Pregnant or lactating woman or without contraception (for child bearing potential women)
* Patient deprived of liberty or under supervision of a guardian
* Impossibility to undergo medical examinations of the study for geographical, social or psychological reasons
* Usual contra-indications for allogenic transplant
* Aged < 55 years
* History of allogenic transplant
* Concomitant neoplastic disease
* Evolutive psychiatric disease
* HIV seropositivity or C hepatitis under treatment
* Women of childbearing age or man, in the absence of effective contraception during treatment and up to 12 months after treatment discontinuation

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2020-03

PRIMARY OUTCOMES:
rates progression free survival 2 years | Time to progression or death

SECONDARY OUTCOMES:
Plasmatic concentration of Busulfan | Time from inclusion until Day -1 before allogenic transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr